CLINICAL TRIAL: NCT03989453
Title: Physical Activity, Menopause and Health. Effects of 12-week Chi Kung Program
Brief Title: Effects of Chi Kung to Improve the Symptoms of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University-Jaén
Record Dates: First submitted 2019-06-04; First posted 2019-06-18 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Quality of Life and Menopause

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment to the groups will be of simple random type and hidden. Those responsible for admitting patients to the intervention phase will not know what group has been assigned each. This assignment will be made in advance by a researcher who will not intervene in the later stages of evaluation, intervention, data recording and elaboration of database. The assignment will be communicated through sealed and totally opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chi Kung group (Experimental): This group receives physical training based on Chi Kung.
  Interventions: Other: Chi Kung
- Control Group (No Intervention): This group does not receive any treatment.

INTERVENTIONS:
Other: Chi Kung — The duration of the intervention is 12 weeks, with 2 sessions per week of Chi Kung. Each session lasts approximately 1 hour and is structured in three parts: initial warm-up (Based on breathing and concentration exercises), of 10 minutes duration, a 40-45 minute Chi Kung session and finally 10 minutes of guided relaxation.
  Arms: Chi Kung group

SUMMARY:
To analyze the effects of a Chi Kung exercise program in Spanish menopausal women

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 2 arms (Control group and experimental group), in which a pre-treatment-postest design has been used.

The study will define two groups:

A control group (CG) that will not be submitted to treatment, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity and will be given a guide to recommendations for promoting physical activity.

An experimental group (GE) that after an initial evaluation will undergo a physical training program based on Chi Kung exercises.

Once the intervention is finished, it will be submitted to a final evaluation to see if there is a difference or not with the results obtained at the beginning.

ELIGIBILITY:
Inclusion Criteria:

* Cessation of menstrual activity for twelve months or more.
* Being able to understand the instructions and exercise protocols of this project

Exclusion Criteria:

* Contraindications for the performance of physical tests, cancer or serious illness, musculoskeletal and neurological diseases, taking of drugs that affect the central nervous system or antidepressants, or lack of will to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 117 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
PSQI (Pittsburgh Sleep Quality Index) | At the beginning-at three months
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result.
STABILOMETRIC PLATFORM | At the beginning-at three months
  instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions
WHQ (The Women's Health Questionnaire) | At the beginning-at three months
  Measures the quality of life related to health specific for menopause
FSFI (The Female Sexual Function Index) | At the beginning-at three months
  Questionnaire that evaluates the sexuality of women during the last four weeks.
MRS (Menopause Rating Scale) | At the beginning-at three months
  Assesses the severity of menopause-related complaints and the impact on health-related quality of life. Calculated by adding up the 11 questions in the questionnaire. Each item has a score of 0-1-2-3-4, with 4 being the worst score.
ABC-16 (Activities Specific Balance Confidence Scale) | At the beginning-at three months
  Questionnaire that assesses balance confidence in performing activities of daily living. It is calculated by adding up the 16 responses of the questionnaire, with 0 being the minimum score and 100 being the maximum score. The higher value represents a better result.

SECONDARY OUTCOMES:
Handgrip Strength | At the beginning-at three months.
  Dynamometer will be employed to assess handgrip strength.
HADS (The Hospital Anxiety And Depression) | At the beginning-at three months.
  A reliable, valid and practical screening tool for identifying and quantifying anxiety and/or depression in non-patients.
SF-36 (The Short Form-36 Health Survey) | At the beginning-at three months.
  Used extensively for assessing health-related quality of life.
TUG (Timed Up and Go test) | At the beginning-at three months.
  Is a simple test used to assess a person's mobility and physical function
BMI (Body Mass Index) | At the beginning-at three months.
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat
Waist circumference | At the beginning-at three months.
  Is used to assess central fat distribution and degree of abdominal obesity.
Waist-to-hip ratio | At the beginning-at three months.
  Is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement.
Cervantes Scale | At the beginning-at three months.
  Specific Scale for better quality of life related to specific health for menopause.
The Female Genital Self-Image Scale (FGSIS) | At the beginning-at three months.
  Scale that evaluates the degree of satisfaction of their own genitals.
FSS (Fatigue Severity Scale) | At the beginning-at three months.
  A self-report scale describing the severity of fatigue and the impact of fatigue on activities of daily living.
FES-I (Falls Efficacy Scale-International) | At the beginning-at three months.
  Questionnaire that evaluates the fear of falling.

CONTACTS AND LOCATIONS:
Locations (1):
- U.E.D. Virgen de la Capilla, Jaén, Spain

REFERENCES:
- [Derived] Carcelen-Fraile MDC, Aibar-Almazan A, Martinez-Amat A, Jimenez-Garcia JD, Brandao-Loureiro V, Garcia-Garro PA, Fabrega-Cuadros R, Rivas-Campo Y, Hita-Contreras F. Qigong for mental health and sleep quality in postmenopausal women: A randomized controlled trial. Medicine (Baltimore). 2022 Sep 30;101(39):e30897. doi: 10.1097/MD.0000000000030897. PMID 36181076
- [Derived] Carcelen-Fraile MDC, Hita-Contreras F, Martinez-Amat A, Loureiro VB, Loureiro NEM, Jimenez-Garcia JD, Fabrega-Cuadros R, Aibar-Almazan A. Impact of Qigong exercises on the severity of the menopausal symptoms and health-related quality of life: A randomised controlled trial. Eur J Sport Sci. 2023 Apr;23(4):656-664. doi: 10.1080/17461391.2022.2044915. Epub 2022 Mar 7. PMID 35179431
- [Derived] Carcelen-Fraile MDC, Aibar-Almazan A, Martinez-Amat A, Brandao-Loureiro V, Jimenez-Garcia JD, Castellote-Caballero Y, Hita-Contreras F. Qigong for Muscle Strength and Static Postural Control in Middle-Aged and Older Postmenopausal Women: A Randomized Controlled Trial. Front Med (Lausanne). 2021 Dec 8;8:784320. doi: 10.3389/fmed.2021.784320. eCollection 2021. PMID 34957157